CLINICAL TRIAL: NCT02348489
Title: A Phase 3, Multicenter, Open-label, Randomized Study of SGI-110 Versus Treatment Choice (TC) in Adults With Previously Untreated Acute Myeloid Leukemia (AML) Who Are Not Considered Candidates for Intensive Remission Induction Chemotherapy
Brief Title: SGI-110 in Adults With Untreated Acute Myeloid Leukemia (AML), Not Considered Candidates for Intensive Remission Induction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGI-110-04
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: AML; Acute Myeloid Leukemia; SGI-110; DNA Hypomethylating Agen
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SGI-110 (guadecitabine) (Experimental): Guadecitabine 60 mg/m^2 administered subcutaneously (SC) daily for 5 days (Days 1-5) in 28-day cycles.
  Interventions: Drug: SGI-110 (guadecitabine)
- Treatment Choice (Active Comparator): One of the following treatment regimens: 20 mg cytarabine administered subcutaneously (SC) twice daily (BID) on Days 1-10 every 28 days; 20 mg/m^2 decitabine given as a 1-hour intravenous (IV) infusion daily on Days 1-5 every 28 days; or 75 mg/m^2 azacitidine given IV or SC daily on Days 1-7 every 28 days.
  Interventions: Drug: Treatment Choice

INTERVENTIONS:
Drug: SGI-110 (guadecitabine) — Investigational medicinal product
  Arms: SGI-110 (guadecitabine)
Drug: Treatment Choice — Choice of one: cytarabine, decitabine, or azacitidine
  Arms: Treatment Choice

SUMMARY:
To compare efficacy and safety between SGI-110 and Treatment Choice in adults with previously untreated AML who are not considered candidates for intensive remission induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Cytologically or histologically confirmed diagnosis of AML (except M3 acute promyelocytic leukemia) according to World Health Organization (WHO) classification.

Performance status (ECOG) of 0-3. Adults with previously untreated AML except for hydroxyurea or corticosteroids. Prior hydroxyurea or lenalidomide treatment for myelodysplastic syndrome (MDS) is allowed.

Not considered candidates for intensive remission induction chemotherapy at time of enrollment based on EITHER:

1. ≥75 years of age OR
2. <75 years of age with at least 1 of the following:

i. Poor performance status (ECOG) score of 2-3.

ii. Clinically significant heart or lung comorbidities, as reflected by at least 1 of:

1. Left ventricular ejection fraction (LVEF) ≤50%.
2. Lung diffusing capacity for carbon monoxide (DLCO) ≤65% of expected.
3. Forced expiratory volume in 1 second (FEV1) ≤65% of expected.
4. Chronic stable angina or congestive heart failure controlled with medication.

iii. Liver transaminases >3 × upper limit of normal (ULN).

iv. Other contraindication(s) to anthracycline therapy (must be documented).

v. Other comorbidity the investigator judges incompatible with intensive remission induction chemotherapy, which must be documented and approved by the study medical monitor before randomization.

Creatinine clearance as estimated by the Cockcroft-Gault (C-G) or other medically acceptable formulas ≥30 mL/min.

Exclusion Criteria:

Candidate for intensive remission induction chemotherapy at the time of enrollment.

Candidate for best supportive care only, ie, not a candidate for any active therapy with the TC comparators.

Known extramedullary central nervous system (CNS) AML.

Second malignancy currently requiring active therapy except breast or prostate cancer stable on or responding to endocrine therapy.

Prior treatment with decitabine or azacitidine.

Hypersensitivity to decitabine, SGI-110, or SGI-110 excipients.

Known active human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection. Inactive hepatitis carrier status or low viral hepatitis titer on antivirals is allowed.

Known significant mental illness or other condition such as active alcohol or other substance abuse or addiction that, in the opinion of the investigator, predisposes the subject to high risk of noncompliance with the protocol.

Refractory congestive heart failure unresponsive to medical treatment; active infection resistant to all antibiotics; or advanced pulmonary disease requiring >2 liters per minute (LPM) oxygen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 815 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-06-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (135):
- United States (23):
  - Mayo Clinic Cancer Center, Scottsdale, Arizona
  - Scripps Cancer Center, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Westwood, Kansas
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - John Theurer Cancer Center at Hackensack, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke Cancer Center, Durham, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University Hospitals Monarch Medical Center, Cleveland, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
- Austria (2):
  - Medizinische Universität Graz, Graz, Styria
  - Hanusch Krankenhaus Wiener Gebietskrankenkasse, Vienna, Vienna
- Belgium (3):
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - UZ Gent, Ghent, Oost-vlaanderen
  - Algemeen Ziekenhuis Sint-Jan, Bruges, West-vlaanderen
- Bulgaria (2):
  - UMHAT 'Sveti Georgi' EAD, Plovdiv
  - Multiprofile Hospital for Active Treatment "Sveta Marina'' EAD, Varna
- Canada (6):
  - Tom Baker Cancer Center, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- Czechia (3):
  - Fakultní nemocnice Brno, Brno, Jihormoravsky KRAJ
  - Všeobecná fakultní nemocnice v Praze, Prague, Prague
  - Fakultní nemocnice Královské Vinohrady, Prague
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet-Copenhagen University Hospital, Copenhagen
  - Odense University Hospital, Odense
- Finland (2):
  - Tampere University Hospital, Tampere, Southern Finland
  - Helsinki University Central Hospital, Helsinki
- France (12):
  - GHR Mulhouse Sud-Alsace, Mulhouse, Alsace
  - Hôpital Hôtel-Dieu, Bayonne, Aquitaine
  - Centre Hospitalier Universitaire Grenoble, La Tronche, Auvergne-Rhône-Alpes
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Centre Henri-Becquerel, Rouen, Haute-normandie
  - CHRU de Limoges - Hôpital Dupuytren, Limoges, Limousin, Lorraine
  - Centre Hospitalier Universitaire de Toulouse, Toulouse, Midi-pyrenees
  - Hôpital Hôtel-Dieu, Nantes, Pays de la Loire Region
  - Institut Paoli Calmettes, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Antoine Lacassagne, Nice, Provence-Alpes-Côte d'Azur Region
  - Hôpital Saint Louis, Paris, Île-de-France Region
- Germany (7):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen, Baden-Wurttemberg
  - Universitätsklinikum Frankfurt Goethe Universität, Frankfurt am Main, Hesse
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig, Lower Saxony
  - Marien Hospital Düsseldorf GmbH, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
- Hungary (4):
  - Bacs-Kiskun Megyei Korhaz, Kecskemét, Bács-Kiskun county
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
- Italy (13):
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro, Pesaro E Urbino
  - IRCCS Centro di Riferimento Oncologico di Basilicata di Rionero in Vulture, Rionero in Vulture, Potenza
  - Azienda Ospedaliero-Univesitaria San Luigi Gonzaga, Orbassano, Torino
  - Azienda Ospedaliera SS. Antonio E. Biagio E. Cesare Arrigo di Alessandria, Alessandria
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Ospedale di Busto Arsizio, Busto Arsizio
  - Azienda Ospedaliera-Universitaria Vittorio Emanuele-Ferrarotto-Santo Bambino, Catania
  - IRCCS Azienda Ospedaliera Universitaria San Martino - IST, Genova
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena
  - AORN A. Cardarelli, Napoli
  - Azienda Policlinico Umberto I di Roma, Roma
  - Azienda Ospedaliero Universitaria S. Maria della Misericordia di Udine, Udine
- Japan (6):
  - Chugoku
  - Chūbu
  - Kanto
  - Kinki
  - Kyushu
  - Tōhoku
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Poland (7):
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin, Lublin Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw, Masovian Voivodeship
  - Szpital Wojewódzki w Opolu - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Opole, Opole Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespól Szpitali Miejskich, Chorzów, Silesian Voivodeship
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Lódz, Łódź Voivodeship
- Romania (2):
  - Spitalul Clinic Judetean de Urgenta Tirgu-Mures, Târgu Mureş, Mureș County
  - Institutul Regional de Oncologie Iasi, Iași
- Russia (3):
  - Ryazan Regional Clinical Hospital, Ryazan
  - Saratov State Medical University, Saratov
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Clinical Centre of Vojvodina, Novi Sad
- South Korea (10):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Seoul National University Hospital, Jongno Gu, Seoul
  - Inje University Busan Paik Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (10):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Vall d´Hebrón, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital General Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Sweden (2):
  - Skånes Universitetssjukhus i Lund, Lund, Skåne County
  - Karolinska University Hospital Huddinge, Stockholm
- Taiwan (5):
  - Chang Gung Medical Foundation-LinKou Branch, Taoyuan District, Taoyuan
  - China Medical University Hospital, Taichung
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (3):
  - Chelsea and Westminster Hospital NHS Foundation Trust, London, England
  - King's College Hospital, London, England
  - Medway Maritime Hospital, Gillingham, Kent

REFERENCES:
- [Derived] Fenaux P, Gobbi M, Kropf PL, Issa JJ, Roboz GJ, Mayer J, Krauter J, Robak T, Kantarjian H, Novak J, Jedrzejczak WW, Thomas X, Ojeda-Uribe M, Miyazaki Y, Min YH, Yeh SP, Brandwein J, Gercheva-Kyuchukova L, Demeter J, Griffiths E, Yee K, Dohner K, Hao Y, Keer H, Azab M, Dohner H. Guadecitabine vs treatment choice in newly diagnosed acute myeloid leukemia: a global phase 3 randomized study. Blood Adv. 2023 Sep 12;7(17):5027-5037. doi: 10.1182/bloodadvances.2023010179. PMID 37276510

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 949 participants were assessed for inclusion in the study. Of these, 134 participants failed screening assessments and 815 participants were randomized.
Pre-assignment Details: For the efficacy analysis (all randomized participants), the total duration was 38 months, with a median follow-up of 766 days (25.5 months), lower quartile follow-up of 671 days (22.4 months), and upper quartile follow-up of 896 days (29.9 months). For safety analysis (all treated participants), total duration was 51 months. Combining participants into a single group as part of the Treatment Choice arm was pre-specified as part of the study design.
Groups:
- SGI-110 (Guadecitabine): Guadecitabine 60 mg/m^2 was administered subcutaneously (SC) daily for 5 days (Days 1-5) in 28-day cycles.
- Treatment Choice: One of the following treatment regimens was administered: 20 mg cytarabine subcutaneously (SC) twice daily (BID) on Days 1-10 every 28 days; 20 mg/m^2 decitabine given as a 1-hour intravenous (IV) infusion daily on Days 1-5 every 28 days; or 75 mg/m^2 azacitidine given IV or SC daily on Days 1-7 every 28 days.
Period: Overall Study
Arm/Group | SGI-110 (Guadecitabine) | Treatment Choice
Started | 408 | 407
Completed | 55 | 40
Not Completed | 353 | 367
Not completed — Death | 336 | 335
Not completed — Withdrawal by Subject | 14 | 27
Not completed — Lost to Follow-up | 3 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Treatment Choice: One of the following treatment regimens was administered: 20 mg cytarabine subcutaneously (SC) BID on Days 1-10 every 28 days; 20 mg/m^2 decitabine given as a 1-hour intravenous (IV) infusion daily on Days 1-5 every 28 days; or 75 mg/m^2 azacitidine given IV or SC daily on Days 1-7 every 28 days.
- Total: Total of all reporting groups
Arm/Group | SGI-110 (Guadecitabine) | Treatment Choice | Total
Number analyzed (Participants) | 408 | 407 | 815
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.9 (6.2) | 75.9 (5.8) | 75.9 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 165 | 342
  Male | 231 | 242 | 473
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 14 | 29
  Not Hispanic or Latino | 365 | 345 | 710
  Unknown or Not Reported | 28 | 48 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 71 | 74 | 145
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 9 | 5 | 14
  White | 311 | 291 | 602
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 15 | 35 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete Response (CR)
Description: Number of participants with a best response of CR assessed based on International Working Group 2003 acute myeloid leukemia (AML) response criteria by a blinded independent pathologist.
Time Frame: Up to 38 months (median follow-up of 25.5 months)
Population: The efficacy analysis set includes all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | SGI-110 (Guadecitabine) | Treatment Choice
Number analyzed (Participants) | 408 | 407
Participants | 79 | 71
Statistical Analysis 1: Comparison: SGI-110 (Guadecitabine) vs Treatment Choice; The complete response rate was compared between the treatment groups using a Cochran Mantel-Haenszel (CMH) test at an alpha level of 0.04 stratified to adjust for stratification factors used at randomization: age (<75 or >=75), Eastern Cooperative Oncology Group (ECOG) performance status (0-1, 2-3), study center region (North American, Europe, Rest of World), and secondary AML (secondary to MDS or other antecedent hematologic disorder) or poor-risk cytogenetics (Yes, No/Unknown); Test type: Superiority; p = 0.482, Cochran-Mantel-Haenszel; Difference in response rate (%) = 1.92, 96% CI 2-sided [-3.67 to 7.5]

2. Primary Outcome: Overall Survival
Description: Survival time was defined as the number of days from the day the participant was randomly assigned to study treatment to the date of death, regardless of cause.
Time Frame: At 676 death events (up to 38 months)
Population: The efficacy analysis set includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | SGI-110 (Guadecitabine) | Treatment Choice
Number analyzed (Participants) | 408 | 407
days | 213 [187 to 255] | 254 [223 to 282]
Statistical Analysis 1: Comparison: SGI-110 (Guadecitabine) vs Treatment Choice; Overall survival curves were estimated using Kaplan-Meier method and compared between the treatment groups using a 2-sided stratification log-rank test, stratified by the same factors used at randomization: age (<75 or >=75), Eastern Cooperative Oncology Group (ECOG) performance status (0-1, 2-3), study center region (North American, Europe, Rest of World), and secondary AML (secondary to MDS or other antecedent hematologic disorder) or poor-risk cytogenetics (Yes, No/Unknown); Test type: Superiority; p = 0.7328, Stratified log-rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.83 to 1.14]

3. Secondary Outcome: Number of Participants With Composite CR (CRc)
Description: CRc is reported as the number of participants with a best response of CR, complete response with incomplete platelet recovery (CRp), or complete response with incomplete blood count recovery (CRi).
Time Frame: Up to 38 months (median follow-up of 25.5 months)
Population: The efficacy analysis set includes all randomized participants.
Measure: Count of Participants; unit: Participants
Groups:
- SGI-110 (Guadecitabine): Guadecitabine 60 mg/m^2 was administered subcutaneously daily for 5 days (Days 1-5) in 28-day cycles.
- Treatment Choice: One of the following treatment regimens were administered: 20 mg cytarabine subcutaneously (SC) BID on Days 1-10 every 28 days; 20 mg/m^2 decitabine given as a 1-hour intravenous (IV) infusion daily on Days 1-5 every 28 days; or 75 mg/m^2 azacitidine given IV or SC daily on Days 1-7 every 28 days.
Arm/Group | SGI-110 (Guadecitabine) | Treatment Choice
Number analyzed (Participants) | 408 | 407
Participants | 93 | 91

4. Secondary Outcome: Number of Days Alive and Out of the Hospital
Description: The date of each hospital admission and discharge was collected for each participant for up to 6 months, unless the participant died or withdrew consent prior to that time. Duration of each hospital stay in days was calculated as date of discharge minus date of admission. The Number of Days Alive and Out of the Hospital (NDAOH) was calculated as: NDAOH=180 - total duration of all hospital stays within 180 days from the first treatment - number of death days before Day 180. For subjects who were lost to follow-up within 6 months, the NDAOH was calculated conservatively assuming that the subject would have died the day after the last contact day.
Time Frame: Month 6
Population: The efficacy analysis set includes all randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | SGI-110 (Guadecitabine) | Treatment Choice
Number analyzed (Participants) | 408 | 407
days | 98.1 (63.6) | 105.7 (63.58)

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the number of days from randomization to the earliest date of investigator's assessment of disease progression, participant receiving an alternative anti-leukemia therapy (including hematopoietic cell transplant), or relapse by peripheral blood (PB) assessment or blinded bone marrow (BM) assessment, whichever occurred first, or death, regardless of cause.
Time Frame: Up to 38 months (median follow-up of 25.5 months)
Population: The efficacy analysis set includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | SGI-110 (Guadecitabine) | Treatment Choice
Number analyzed (Participants) | 408 | 407
days | 159 [136 to 178] | 166 [148 to 179]

6. Secondary Outcome: Number of Red Blood Cell or Platelet Transfusions
Description: The total number of red blood cells (RBCs) transfused or, separately, the total number of platelets transfused up to the 6-month time point for each participant was counted from the date of randomization to Day 180, the date of last contact, or date of death, whichever occurred earlier. One RBC or platelet transfusion was defined as one unit, and a single bag of RBCs or platelets was considered one unit.
Time Frame: Month 6
Population: The efficacy analysis set includes all randomized participants.
Measure: Mean (Standard Deviation); unit: transfusion units
Arm/Group | SGI-110 (Guadecitabine) | Treatment Choice
Number analyzed (Participants) | 408 | 407
transfusion units
  Red Blood Cell Transfusions | 16.2 (11.84) | 15.6 (13.02)
  Platelet Transfusions | 12.5 (18.78) | 14.4 (39.10)

7. Secondary Outcome: Change in Health-related Quality of Life (QOL) Scores From Baseline: EQ-5D-5L
Description: EuroQol 5-level 5-dimension (EQ-5D-5L) descriptive scores were collected for each participant for a minimum of 6 months, unless the participant died or withdrew consent. Scores within each dimension for EQ-5D (mobility, self-care, usual activity, pain/discomfort, anxiety/depression) were calculated using counts and proportions. Mean change in scores from baseline are summarized in which an index score of 0 represents the worst health state and 1 represents the best health state.
Time Frame: Baseline to Month 6
Population: The efficacy analysis set includes all randomized participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SGI-110 (Guadecitabine) | Treatment Choice
Number analyzed (Participants) | 391 | 378
score on a scale
  Baseline | 0.7767 (0.2160) | 0.7663 (0.2291)
  Month 6: number analyzed (Participants) | 180 | 183
  Month 6 | 0.8252 (0.1825) | 0.8240 (0.1948)
  Change from Baseline: number analyzed (Participants) | 177 | 178
  Change from Baseline | -0.0023 (0.1830) | 0.0112 (0.2325)

8. Secondary Outcome: Change in Health-related Quality of Life (QOL) Scores From Baseline: EQ-VAS
Description: EuroQol-Visual Analogue Scale (EQ-VAS) descriptive scores were collected for each participant for a minimum of 6 months, unless the participant died or withdrew consent. A vertical 20-cm scale for EQ-VAS was used where the lowest value of 0 was labeled "the worst health you can imagine" and the top value of 100 was labeled "the best health you can imagine." Mean change in scores from baseline are summarized.
Time Frame: Baseline to Month 6
Population: The efficacy analysis set includes all randomized participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SGI-110 (Guadecitabine) | Treatment Choice
Number analyzed (Participants) | 391 | 377
score on a scale
  Baseline | 64.64 (21.69) | 63.58 (21.05)
  Month 6: number analyzed (Participants) | 180 | 183
  Month 6 | 72.76 (18.61) | 71.72 (18.88)
  Change from Baseline: number analyzed (Participants) | 177 | 178
  Change from Baseline | 3.28 (19.35) | 3.67 (22.16)

9. Secondary Outcome: Duration of CR
Description: Duration of CR (in number of days) was calculated from the first time a CR was observed to the time of relapse, defined as the earliest time point whereby BM assessment or PB assessment indicated relapse/disease progression due to reappearance of leukemic blasts in PB or ≥ 5% leukemic blasts in BM.
Time Frame: Up to 38 months (median follow-up of 25.5 months)
Population: The efficacy analysis set includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | SGI-110 (Guadecitabine) | Treatment Choice
Number analyzed (Participants) | 408 | 407
days | 217 [175 to 261] | 231 [182 to 289]

ADVERSE EVENTS:
Time Frame: Up to 51 months. Median (range) duration of treatment was 5 cycles (1-42) for SGI-110 and 5 cycles (1-37) for Treatment Choice (28 days per cycle). Treatment-emergent adverse events were events that first occurred or worsened after the first dose of study treatment until 30 days after the last dose or start of an alternative anti-leukemia treatment, whichever occurred first.
Description: Safety analysis set (randomized participants who received study treatment) was analyzed for TEAEs. All-cause mortality is presented for all randomized participants (participant flow shows number of deaths with primary reason for study withdrawal). Combining participants into a single group (Treatment Choice) was pre-specified as part of the study design and data for each treatment in that arm were not analyzed separately. Death is listed as an SAE when there is no identifiable cause or event.
Arm/Group | SGI-110 (Guadecitabine) | Treatment Choice
All-Cause Mortality (participants affected / at risk) | 341/408 | 344/407
Serious Adverse Events (participants affected / at risk) | 327/401 | 297/392
Other Adverse Events (participants affected / at risk) | 379/401 | 371/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SGI-110 (Guadecitabine) (N=401) | Treatment Choice (N=392)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 101 (147) | 88 (138)
Hemorrhagic diathesis (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Histiocytosis hematophagic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 6 (7) | 2 (2)
Lymphoadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphoadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Monoclonal B-cell lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (15) | 5 (5)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (6) | 3 (3)
Angina pectoris (Cardiac disorders) | 3 (4) | 4 (4)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 6 (13)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3) | 9 (9)
Cardiac failure (Cardiac disorders) | 8 (8) | 10 (11)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 4 (7) | 3 (3)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Mastoid disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 1 (2) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (4) | 2 (2)
Colitis ischemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 8 (9) | 7 (10)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (3) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 3 (3) | 2 (2)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 4 (4)
Small intestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (2)
Asthenia (General disorders) | 2 (2) | 4 (4)
Catheter site erythema (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 5 (5) | 5 (5)
Device related thrombosis (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 9 (9) | 10 (10)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 5 (5) | 4 (4)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Edema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 16 (19) | 13 (14)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (2)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (2) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 3 (3) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 3 (3) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Bacteremia (Infections and infestations) | 7 (8) | 2 (2)
Bacterial infection (Infections and infestations) | 2 (2) | 1 (1)
Bacteroides bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 6 (6) | 2 (2)
Bronchopulmonary aspergillosis (Infections and infestations) | 2 (2) | 2 (2)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 3 (4) | 6 (7)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 1 (1)
Clostridium colitis (Infections and infestations) | 1 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 4 (4) | 2 (3)
Clostridium difficile infection (Infections and infestations) | 4 (5) | 2 (2)
Cystitis (Infections and infestations) | 3 (3) | 0 (0)
Dermo-hypodermitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 4 (4) | 7 (8)
Device related sepsis (Infections and infestations) | 2 (2) | 2 (2)
Diverticulitis (Infections and infestations) | 4 (6) | 1 (1)
Encephalomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 2 (2)
Escherichia bacteremia (Infections and infestations) | 2 (2) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis pseudomonas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1)
Hematoma infection (Infections and infestations) | 2 (2) | 0 (0)
Hepatosplenic abscess (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster oticus (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 6 (6) | 5 (6)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 6 (6) | 3 (3)
Injection site abscess (Infections and infestations) | 1 (1) | 0 (0)
Injection site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 3 (3) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Localized infection (Infections and infestations) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Mucormycosis (Infections and infestations) | 1 (1) | 1 (1)
Muscle abscess (Infections and infestations) | 1 (1) | 1 (1)
Neutropenic infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 1 (1)
Parotitis (Infections and infestations) | 2 (3) | 0 (0)
Pathogen resistance (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Periumbilical abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (2)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 117 (147) | 79 (102)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 62 (83) | 44 (58)
Septic shock (Infections and infestations) | 16 (17) | 17 (19)
Septic vasculitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 4 (4)
Sinusitis fungal (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 3 (3) | 2 (2)
Staphylococcal bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 3 (3)
Streptococcal bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1)
Systemic infection (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 2 (3) | 1 (1)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Urethritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 14 (16) | 10 (11)
Urinary tract infection enterococcal (Infections and infestations) | 3 (3) | 0 (0)
Urosepsis (Infections and infestations) | 3 (3) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 2 (2) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subarachnoid hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Subdural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 3 (3) | 3 (3)
Influenza A virus test positive (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 4 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle hemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumor associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 1 (1) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 6 (6) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhage intracranial (Nervous system disorders) | 1 (1) | 4 (5)
Hemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial hematoma (Nervous system disorders) | 0 (0) | 1 (1)
Ischemic stroke (Nervous system disorders) | 2 (2) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (2)
Seizure (Nervous system disorders) | 2 (2) | 2 (2)
Syncope (Nervous system disorders) | 2 (2) | 4 (6)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 2 (2)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 4 (4) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 11 (11) | 15 (16)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis hemorrhagic (Renal and urinary disorders) | 1 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4) | 2 (2)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Rash generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 5 (5) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 3 (3) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 3 (3)
Iliac artery embolism (Vascular disorders) | 0 (0) | 1 (1)
Leriche syndrome (Vascular disorders) | 1 (1) | 0 (0)
Lupus vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shock hemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 2 (2) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SGI-110 (Guadecitabine) (N=401) | Treatment Choice (N=392)
Anemia (Blood and lymphatic system disorders) | 88 (211) | 78 (201)
Febrile neutropenia (Blood and lymphatic system disorders) | 66 (103) | 40 (57)
Leukopenia (Blood and lymphatic system disorders) | 37 (120) | 33 (124)
Neutropenia (Blood and lymphatic system disorders) | 115 (319) | 88 (233)
Thrombocytopenia (Blood and lymphatic system disorders) | 116 (380) | 101 (313)
Abdominal pain (Gastrointestinal disorders) | 30 (43) | 46 (50)
Abdominal pain upper (Gastrointestinal disorders) | 21 (25) | 15 (16)
Constipation (Gastrointestinal disorders) | 125 (166) | 114 (168)
Diarrhea (Gastrointestinal disorders) | 122 (169) | 83 (116)
Hemorrhoids (Gastrointestinal disorders) | 24 (28) | 19 (24)
Nausea (Gastrointestinal disorders) | 91 (141) | 108 (150)
Stomatitis (Gastrointestinal disorders) | 46 (59) | 38 (44)
Vomiting (Gastrointestinal disorders) | 58 (80) | 66 (82)
Asthenia (General disorders) | 61 (102) | 55 (81)
Fatigue (General disorders) | 63 (97) | 50 (74)
Injection site reaction (General disorders) | 73 (148) | 48 (75)
Edema peripheral (General disorders) | 95 (125) | 78 (108)
Pain (General disorders) | 21 (22) | 14 (14)
Pyrexia (General disorders) | 89 (155) | 110 (176)
Bronchitis (Infections and infestations) | 22 (30) | 13 (15)
Cellulitis (Infections and infestations) | 29 (37) | 22 (25)
Nasopharyngitis (Infections and infestations) | 18 (27) | 20 (21)
Oral candidiasis (Infections and infestations) | 23 (27) | 17 (21)
Oral herpes (Infections and infestations) | 31 (36) | 20 (21)
Pneumonia (Infections and infestations) | 54 (64) | 31 (34)
Upper respiratory tract infection (Infections and infestations) | 22 (34) | 20 (28)
Urinary tract infection (Infections and infestations) | 33 (46) | 28 (39)
Contusion (Injury, poisoning and procedural complications) | 20 (23) | 22 (27)
Fall (Injury, poisoning and procedural complications) | 34 (43) | 29 (37)
Weight decreased (Investigations) | 35 (47) | 25 (28)
Decreased appetite (Metabolism and nutrition disorders) | 89 (116) | 62 (80)
Hyperkalemia (Metabolism and nutrition disorders) | 24 (33) | 13 (19)
Hypoalbuminemia (Metabolism and nutrition disorders) | 26 (36) | 23 (43)
Hypocalcemia (Metabolism and nutrition disorders) | 25 (30) | 18 (29)
Hypokalemia (Metabolism and nutrition disorders) | 96 (173) | 77 (128)
Hypomagnesemia (Metabolism and nutrition disorders) | 31 (50) | 27 (36)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (28) | 35 (39)
Back pain (Musculoskeletal and connective tissue disorders) | 34 (43) | 36 (43)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17 (20) | 20 (22)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 40 (51) | 32 (39)
Dizziness (Nervous system disorders) | 36 (47) | 42 (56)
Headache (Nervous system disorders) | 32 (44) | 38 (53)
Anxiety (Psychiatric disorders) | 23 (23) | 22 (24)
Depression (Psychiatric disorders) | 14 (15) | 21 (21)
Insomnia (Psychiatric disorders) | 38 (52) | 45 (56)
Acute kidney injury (Renal and urinary disorders) | 23 (24) | 16 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 79 (100) | 66 (83)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 63 (83) | 51 (60)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 53 (71) | 36 (51)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 (29) | 23 (27)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 21 (23) | 13 (13)
Erythema (Skin and subcutaneous tissue disorders) | 21 (21) | 17 (20)
Pruritis (Skin and subcutaneous tissue disorders) | 22 (28) | 26 (32)
Rash (Skin and subcutaneous tissue disorders) | 41 (55) | 28 (33)
Hematoma (Vascular disorders) | 25 (33) | 19 (29)
Hypertension (Vascular disorders) | 28 (42) | 25 (37)
Hypotension (Vascular disorders) | 31 (40) | 31 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-03-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT02348489/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT02348489/SAP_001.pdf